CLINICAL TRIAL: NCT03085121
Title: A Comparative Study of Femoral Extramedullary and Intramedullary Alignment Systems in Total Knee Arthroplasty
Brief Title: Femoral Extramedullary Versus Intramedullary Alignment Systems in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Qing Jiang, Prof., The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUIWAIXZH
Record Dates: First submitted 2017-03-06; First posted 2017-03-21 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Knee Osteoarthritis
Keywords: extramedullary; intramedullary; total knee arthroplasty (TKA)
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Male Extramedullary (Experimental): In this group, patients are male and femoral extramedullary resection would be used.
  Interventions: Procedure: Distal femoral resection in total knee arthroplasty
- Female Extramedullary (Experimental): In this group, patients are female and femoral extramedullary resection would be used.
  Interventions: Procedure: Distal femoral resection in total knee arthroplasty
- Male Intramedullary (Active Comparator): In this group, patients are male and femoral Intramedullary resection would be used.
  Interventions: Procedure: Distal femoral resection in total knee arthroplasty
- Female Intramedullary (Active Comparator): In this group, patients are female and femoral Intramedullary resection would be used.
  Interventions: Procedure: Distal femoral resection in total knee arthroplasty

INTERVENTIONS:
Procedure: Distal femoral resection in total knee arthroplasty — EM and IM alignment systems are used to make the distal femoral cut in a random order.

SUMMARY:
A prospective study will be performed to compare the clinical outcome after total knee arthroplasty (TKA) using two different alignment systems: an extramedullary system versus an intramedullary system. The extramedullary femoral alignment system is newly designed. These two systems are used to make the distal femoral resection in 100 patients in a random order.

ELIGIBILITY:
Inclusion Criteria:

* Varus knee; degrees of extra articular deformity < 15°; Knee Osteoarthritis; Straight limited < 30°; range of knee flexion > 90°; No hip abnormalities

Exclusion Criteria:

* Valgus knee; degrees of extra articular deformity > 15°; Knee infection; Rheumatic arthritis; Ankylosing Spondylitis; Prior femoral surgery

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-04-04 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Imaging tests | pre surgery and 3, 12 months post surgery
  Evaluate the X-ray changes. Measuring the hip-knee-ankle (HKA) angle by x-ray films
Assess the changes of KSS scores | pre surgery and 3, 12 months post surgery
  KSS scores will be recorded.
Assess the changes of SF-36 scores | pre surgery and 3, 12 months post surgery
  SF-36 scores will be recorded
Assess the changes of WOMAC scores | pre surgery and 3, 12 months post surgery
  WOMAC scores will be recorded.

SECONDARY OUTCOMES:
deep vein thrombosis (DVT) | pre surgery and 3, 12 months post surgery
  DVT was diagnosed by 3 experienced radiologists 96 according to Robinov group's criterion.
Range of knee motion | pre surgery and 3, 12 months post surgery
  Range of knee motion will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhihong Xu, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meding JB, Berend ME, Ritter MA, Galley MR, Malinzak RA. Intramedullary vs extramedullary femoral alignment guides: a 15-year follow-up of survivorship. J Arthroplasty. 2011 Jun;26(4):591-5. doi: 10.1016/j.arth.2010.05.008. PMID 21575792
- [Background] Nakahara H, Matsuda S, Okazaki K, Tashiro Y, Iwamoto Y. Sagittal cutting error changes femoral anteroposterior sizing in total knee arthroplasty. Clin Orthop Relat Res. 2012 Dec;470(12):3560-5. doi: 10.1007/s11999-012-2397-1. Epub 2012 May 19. PMID 22610529
- [Background] Kim CW, Seo SS, Kim JH, Lee HJ, Lee CR. Factors affecting the osteolysis around the components after posterior-stabilized total knee replacement arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2015 Jun;23(6):1863-9. doi: 10.1007/s00167-014-3088-0. Epub 2014 Jun 11. PMID 24912573